CLINICAL TRIAL: NCT05309967
Title: Effect of Glutaraldehyde-based Desensitizer in the Control of Tooth Sensitivity and Tooth Color Post- Whitening : a Randomized, Single Blind and Split Mouth Clinical Trial.
Brief Title: Effect of Glutaraldehyde-based Desensitizer in the Control of Tooth Sensitivity and Tooth Color Post- Whitening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Associate Professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UFpara-0012
Record Dates: First submitted 2022-03-15; First posted 2022-04-04 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Dentin Sensitivity
Keywords: Tooth Bleaching; dentin adhesives; tooth sensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: It is a split mouth study composed of two groups randomized between left and right sides.
Who Masked: Participant, Investigator
Masking Description: For the double-blind study, the evaluator and the patient will be blinded. The bleaching procedure and the therapies under study will be performed by one operator and will only involve one evaluator not participant in the randomization and without knowledge of the interventions applied in the groups. The evaluator will be responsible for measuring and tabulating information regarding sensitivity, color analysis and the impact on patients' quality of life.
  The desensitizer and its placebo will be placed in similar containers so that they cannot be identified by the volunteers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLUMA (Experimental): Glutaraldehyde + Hydroxyethyl methacrylate (GLUMA® Desensitizer)
  Interventions: Other: GLUMA DESINSITIZER
- PLACEBO (Placebo Comparator): DISTILLED WATER
  Interventions: Other: PLACEBO

INTERVENTIONS:
Other: GLUMA DESINSITIZER — GLUTARALDEHYDE
  Arms: GLUMA
Other: PLACEBO — DESTILLED WATER
  Arms: PLACEBO

SUMMARY:
Tooth whitening is one of the most indicated aesthetic procedures in dentistry and there is evidence that it interferes with aspects of patients' quality of life. However, the sensitivity, associated with the post-procedure period, challenges clinicians and researchers. The use of topic desensitizing agents could be a alternative for the control of this adverse effects of bleaching agents. The objective of this randomized clinical study, therefore, is to evaluate the effect of glutaraldehyde-based desensitizing agent associated on tooth sensitivity and tooth color after bleaching with 35% hydrogen peroxide. 25 patients will be selected divided into two groups for a double-blind and split-mouth study. Among the results it is expected: that the use of glutaraldehyde desensitizing agent helps in the control of post-bleaching sensitivity, without harming the final color obtained of patients submitted to the proposed clinical protocol.

DETAILED DESCRIPTION:
Tooth whitening will be performed in 3 sessions with an interval of 7 days. Desensitizing agent and placebo will be applied in all sessions in a split mouth design . All groups will receive in-office bleaching treatment according to the steps described below:1 Prophylaxis; 2- Application of gingival barrier; 3- Application of the desensitizing product or placebo in accordance with the established groups; 4- Handling the bleaching material following the manufacturer's instructions: applications of whiteness HP35% bleaching gel for 15 minutes each, totaling 45 minutes; 5- Final removal of the whitening gel and the gingival barrier followed by washing with water.

Application of the desensitizer or its placebo (step 3) will follow the following sequence:1. Relative insulation with cotton rolls; 2- Active application of the product on the buccal surfaces of all teeth with the aid of a Microbrush for 10 seconds.; 3- Wait 60 seconds and apply a light jet of air until the tooth surface is no longer shiny; 4- Wash with water for 10 seconds.

To assess the patient's perception of pain, participants will be provided with a questionnaire to be filled out daily for 21 days from the first whitening treatment session. The criteria are based on the personal perception of the pain threshold, related to the level of sensitivity caused by bleaching treatment. The visual analogue scale (VAS) will be adopted as a reference. Numerical scale on which the number 0 (zero) corresponds to total absence of pain and 10 (ten) to maximum bearable pain.

The color records of the bleached teeth will be performed by a single evaluator who will do it session :T0- baseline, T1- a week after the first session; T2- a week after the second session; T3- a week after the third session. An area of interest for color registration will be the middle third of the buccal surface of the teeth, following the the guidelines of the American Dental Association. Visual analysis will be performed using a Vita Classical scale following a color scale order organized by value. A second color analysis will be performed with the aid of a spectrophotometer that acts according to the CIELab and CIEDE 2000 system. The region for color evaluation with the Easyshade will be standardized as the middle third of the buccal surface of the anterior teeth.

ELIGIBILITY:
Inclusion Criteria:

* healthy incisors, canines and premolars;
* Do not having a diagnosis of dental hypersensitivity.
* Do not have been at desensitizing treatment in the past two years.
* Do not have been done dental whitening treatment.

Exclusion Criteria:

* Patients undergoing orthodontic treatment;

  * Presence of periodontal disease;
  * Presence of cracks or fractures in the teeth
  * Presence of restorations and prostheses in anterior teeth;
  * Presence of extensive restorations and/or deep in molars;
  * Patients with serious dental darkening internal or external ;
  * Presence of exposed dentin.
  * Pregnant and lactating women.
  * Patients on active treatment whom are using anti-inflammatory drugs and painkillers.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Use of glutaraldehyde based material with or without low level laser therapy in tooth sensitivity during whitening protocol with 35 % hydrogen peroxide. | Patients will be evaluated during 21 days.
  Self-reported pain intensity will be assessed daily, during 21 days, through self-perception questionnaire, answered by the patients from the first tooth bleaching session until one week after the last session. The evaluation will be performed by each patient, according to a numeric visual analog scale, as follows: 0 - 10. Where 0 correspond to no pain and 10 the most severe pain that patient have been ever identified
Use of glutaraldehyde based material with or without low level laser therapy in patient´s quality of life after whitening protocol with 35 % hydrogen peroxide. | 6 months
  A questionnaire will be applied before the bleaching treatment, after the completion of the bleaching treatment and 6 months after bleaching as a follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Raissa Araujo de Mesquita, Belém, Pará, Brazil

REFERENCES:
- [Background] de Paula B, Alencar C, Ortiz M, Couto R, Araujo J, Silva C. Effect of photobiomodulation with low-level laser therapy combined with potassium nitrate on controlling post-bleaching tooth sensitivity: clinical, randomized, controlled, double-blind, and split-mouth study. Clin Oral Investig. 2019 Jun;23(6):2723-2732. doi: 10.1007/s00784-018-2715-4. Epub 2018 Oct 25. PMID 30361793
- [Background] Shulman JD, Maupome G, Clark DC, Levy SM. Perceptions of desirable tooth color among parents, dentists and children. J Am Dent Assoc. 2004 May;135(5):595-604; quiz 654-5. doi: 10.14219/jada.archive.2004.0247. PMID 15202751
- [Background] Alkhatib MN, Holt R, Bedi R. Prevalence of self-assessed tooth discolouration in the United Kingdom. J Dent. 2004 Sep;32(7):561-6. doi: 10.1016/j.jdent.2004.06.002. PMID 15386863
- [Background] Rezende M, Loguercio AD, Kossatz S, Reis A. Predictive factors on the efficacy and risk/intensity of tooth sensitivity of dental bleaching: A multi regression and logistic analysis. J Dent. 2016 Feb;45:1-6. doi: 10.1016/j.jdent.2015.11.003. Epub 2015 Dec 2. PMID 26612623
- [Background] Kwon SR, Wertz PW. Review of the Mechanism of Tooth Whitening. J Esthet Restor Dent. 2015 Sep-Oct;27(5):240-57. doi: 10.1111/jerd.12152. Epub 2015 May 13. PMID 25969131
- [Background] Cardenas AFM, Maran BM, Araujo LCR, de Siqueira FSF, Wambier LM, Gonzaga CC, Loguercio AD, Reis A. Are combined bleaching techniques better than their sole application? A systematic review and meta-analysis. Clin Oral Investig. 2019 Oct;23(10):3673-3689. doi: 10.1007/s00784-019-03042-4. Epub 2019 Aug 29. PMID 31468261
- [Background] Kwon SR, Dawson DV, Schenck DM, Fiegel J, Wertz PW. Spectrophotometric Evaluation of Potassium Nitrate Penetration Into the Pulp Cavity. Oper Dent. 2015 Nov-Dec;40(6):614-21. doi: 10.2341/14-214-L. Epub 2015 Jul 7. PMID 26151563
- [Background] Klaric Sever E, Budimir Z, Cerovac M, Stambuk M, Par M, Negovetic Vranic D, Tarle Z. Clinical and patient reported outcomes of bleaching effectiveness. Acta Odontol Scand. 2018 Jan;76(1):30-38. doi: 10.1080/00016357.2017.1376111. Epub 2017 Sep 11. PMID 28893130
- [Background] Caviedes-Bucheli J, Ariza-Garcia G, Restrepo-Mendez S, Rios-Osorio N, Lombana N, Munoz HR. The effect of tooth bleaching on substance P expression in human dental pulp. J Endod. 2008 Dec;34(12):1462-5. doi: 10.1016/j.joen.2008.09.013. Epub 2008 Oct 31. PMID 19026874
- [Background] Vaz MM, Lopes LG, Cardoso PC, Souza JB, Batista AC, Costa NL, Torres EM, Estrela C. Inflammatory response of human dental pulp to at-home and in-office tooth bleaching. J Appl Oral Sci. 2016 Sep-Oct;24(5):509-517. doi: 10.1590/1678-775720160137. PMID 27812622
- [Background] Marto CM, Baptista Paula A, Nunes T, Pimenta M, Abrantes AM, Pires AS, Laranjo M, Coelho A, Donato H, Botelho MF, Marques Ferreira M, Carrilho E. Evaluation of the efficacy of dentin hypersensitivity treatments-A systematic review and follow-up analysis. J Oral Rehabil. 2019 Oct;46(10):952-990. doi: 10.1111/joor.12842. Epub 2019 Jul 12. PMID 31216069
- [Background] de Melo Alencar C, Castro da Silva R, Nogueira Araujo JL, Silva da Silveira AD, Martins Silva C. A clinical, randomized, double-blind study on the use of toothpastes immediately after at-home tooth bleaching. Am J Dent. 2017 Oct;30(5):267-271. PMID 29178730
- [Background] Moosavi H, Arjmand N, Ahrari F, Zakeri M, Maleknejad F. Effect of low-level laser therapy on tooth sensitivity induced by in-office bleaching. Lasers Med Sci. 2016 May;31(4):713-9. doi: 10.1007/s10103-016-1913-z. Epub 2016 Mar 10. PMID 26964798
- [Background] Pompeu DDS, de Paula BLF, Barros APO, Nunes SC, Carneiro AMP, Araujo JLN, Silva CM. Combination of strontium chloride and photobiomodulation in the control of tooth sensitivity post-bleaching: A split-mouth randomized clinical trial. PLoS One. 2021 Apr 28;16(4):e0250501. doi: 10.1371/journal.pone.0250501. eCollection 2021. PMID 33909659
- [Background] Diniz A, Lima S, Tavarez R, Borges AH, Pinto S, Tonetto MR, Loguercio AD, Bandeca MC. Preventive Use of a Resin-based Desensitizer Containing Glutaraldehyde on Tooth Sensitivity Caused by In-office Bleaching: A Randomized, Single-blind Clinical Trial. Oper Dent. 2018 Sep/Oct;43(5):472-481. doi: 10.2341/17-020-C. Epub 2018 Mar 23. PMID 29570018
- [Background] Lopes AO, de Paula Eduardo C, Aranha ACC. Evaluation of different treatment protocols for dentin hypersensitivity: an 18-month randomized clinical trial. Lasers Med Sci. 2017 Jul;32(5):1023-1030. doi: 10.1007/s10103-017-2203-0. Epub 2017 Apr 8. PMID 28391435
- [Background] Qin C, Xu J, Zhang Y. Spectroscopic investigation of the function of aqueous 2-hydroxyethylmethacrylate/glutaraldehyde solution as a dentin desensitizer. Eur J Oral Sci. 2006 Aug;114(4):354-9. doi: 10.1111/j.1600-0722.2006.00382.x. PMID 16911108
- [Background] Parreiras SO, Szesz AL, Coppla FM, Martini EC, Farago PV, Loguercio AD, Reis A. Effect of an experimental desensitizing agent on reduction of bleaching-induced tooth sensitivity: A triple-blind randomized clinical trial. J Am Dent Assoc. 2018 Apr;149(4):281-290. doi: 10.1016/j.adaj.2017.10.025. Epub 2018 Feb 10. PMID 29439773
- [Background] Wong AH, Cheung CS, McGrath C. Developing a short form of Oral Health Impact Profile (OHIP) for dental aesthetics: OHIP-aesthetic. Community Dent Oral Epidemiol. 2007 Feb;35(1):64-72. doi: 10.1111/j.1600-0528.2007.00330.x. PMID 17244139
- [Background] Pires CP, Ferraz MB, de Abreu MH. Translation into Brazilian Portuguese, cultural adaptation and validation of the oral health impact profile (OHIP-49). Braz Oral Res. 2006 Jul-Sep;20(3):263-8. doi: 10.1590/s1806-83242006000300015. PMID 17119711